CLINICAL TRIAL: NCT01219348
Title: IDO Peptid Vaccination in Combination With Immune Stimulating Agent Aldara and the Adjuvant Montanide, for Treatment of Patients With Locally Advanced or Metastatic Non Small-cell Lung Cancer. A First-in-man Phase I Trial.
Brief Title: IDO Peptid Vaccination for Stage III-IV Non Small-cell Lung Cancer Patients.
Acronym: IDOvaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Prof., MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU 1006 - IDO
Record Dates: First submitted 2010-05-10; First posted 2010-10-13 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: NSCLC; Lung Cancer
Keywords: IDO enzyme; Vaccination trial; Immunotherapy; NSCLC, stage III_IV; Indeolamine 2,3 dioxygenase = IDO
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indeolamine 2,3 deoxygenase (Experimental): To inhibit immune suppression and tolerance, by blocking the IDO enzyme with vaccination against IDO.
  Interventions: Biological: IDO peptide vaccination

INTERVENTIONS:
Biological: IDO peptide vaccination — Vaccination every second week

SUMMARY:
Title: IDO peptid vaccination in combination with immune stimulating agent Aldara and the adjuvant Montanide, for treatment of patients with locally advanced or metastatic non small-cell lung cancer. A first-in-man phase I trial.

Hypothesis: In this trial the investigators assess a new immunotherapeutic strategy targeting the immune inhibiting enzyme, IDO to investigate the potential of vaccination against IDO as a possible anticancer target.

DETAILED DESCRIPTION:
Background: Non small-cell lung cancer (NSCLC) is a common disease with a poor prognosis when locally advanced or metastasized, despite advances in surgery, chemo- and radiation therapy.

In this trial the investigators assess a new immunotherapeutic strategy targeting the immune inhibiting enzyme, IDO to investigate the potential of vaccination against IDO as a possible anticancer target.

IDO has recently been recognized as an important factor in immune regulation and development of immune tolerance in the microenvironment of cancer cells. Cells that represent IDO at their surface are known to inhibit the immune system. IDO expression is seen both in cancer cells and antigen presenting cells. The vaccination against IDO expressing cells is therefore two-sided. The vaccination therapy is thought to block the development of immune tolerance induced by IDO expressing cells. At the same time the investigators aim to stimulate the production of IDO specific T-cells, hence facilitating the elimination of IDO positive tumour cells. The primary end points are safety and toxicity evaluation. Secondary end points are immunological and clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological verified non small cell lung cancer 2. Metastatic or locally advanced incurable stage III-IV NSCLC 3. Patients need to be off chemotherapy treatment 4. Evaluable disease according to RECIST V. 1,1 criteria 5. Patients must be HLA-A2 positive 6. Patients > 18 years old 7. Performance status 0-1 8. Life expectancy of > 3 months 9. Acceptable bone marrow function, defined as

a. White blood cell count > 2,5 * 109 /l b. Neutrophil count> 1,5 * 109 /l c. Platelet count > 75 * 109/l 10. Creatinin measured < 2,5 * upper limit value 11. Acceptable liver function, defined as

1. ASAT < 100 U/L
2. Bilirubin < 30 U/L 12. Women with child-bearing potential must have controlled s-hcg before inclusion 13. Patients must provide written informed concent before inclusion 13. Termination of chemotherapy treatment > 28 days before inclusion

   14. Termination of radiotherapy treatment > 28 days before inclusion

   15. Inclusion at least > 4 weeks after complicated gastric surgery

   -

   Exclusion Criteria:
   1. Other malignancies except from non-melanoma skin cancer in the previous 5 years until study inclusion
   2. Brain metastasis are allowed after radical excision, and if the patient at least 1 month afterwards is not in clinical or radiographic progression
   3. Patients with active gastric ulcer disease; patients taking antacid treatment can be included.
   4. Severe medical condition, severe asthma, severe COLD, severe arteriosclerosis or diabetic disease
   5. Acute or chronic infection (ie. HIV, hepatitis, tuberculosis)
   6. Severe allergic reaction or previous anaphylactic shock
   7. Autoimmune diseases (ie. autoimmune neutropenia/thrombopenia, hæmolytic anaemia, systemic lupus erythematosis, Sjøgrens disease, sclerodermia, Goodpastures syndrome, Addisons disease, active Graves disease)
   8. Pregnant or lactating women
   9. Psychiatric disease, which can influence compliance
   10. Known hypersensitivity towards the adjuvance Montanide, the Aldara creme, or adhesive tape.
   11. Treatment with immunosuppressive therapy (ie. dexamethasone, methotrexate)
   12. Treatment with other experimental therapy
   13. Treatment with other anti-cancer therapy, except from treatment of osteoporosis
   14. No systemic chemotherapy, immunotherapy or radiation therapy (except locally) are allowed until 28 days before inclusion.

       -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
evidence of toxicity | 12 months
  CTCAE = Common Terminology Criteria for Adverse Events v. 3.0 will be used for registration of toxicity

SECONDARY OUTCOMES:
evaluation of immunological and clinical responses | 18 months
  immunological assays will be used to identify immunological responses. CT scans will be used for evaluation of clinical responses.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Zeeberg Iversen, MD, Principal Investigator — Center for Cancer Immune Therapy
Locations (2):
- Denmark (2):
  - Center for Cancer ImmuneTherapy, Herlev, Copenhagen
  - Center for Cancer Immune Therapy, Dept. og Haematology/Oncology, Copenhagen, Herlev, Copenhagen

REFERENCES:
- [Derived] Iversen TZ, Engell-Noerregaard L, Ellebaek E, Andersen R, Larsen SK, Bjoern J, Zeyher C, Gouttefangeas C, Thomsen BM, Holm B, Thor Straten P, Mellemgaard A, Andersen MH, Svane IM. Long-lasting disease stabilization in the absence of toxicity in metastatic lung cancer patients vaccinated with an epitope derived from indoleamine 2,3 dioxygenase. Clin Cancer Res. 2014 Jan 1;20(1):221-32. doi: 10.1158/1078-0432.CCR-13-1560. Epub 2013 Nov 11. PMID 24218513
- [Derived] Andersen MH. The specific targeting of immune regulation: T-cell responses against Indoleamine 2,3-dioxygenase. Cancer Immunol Immunother. 2012 Aug;61(8):1289-97. doi: 10.1007/s00262-012-1234-4. Epub 2012 Mar 3. PMID 22388712